CLINICAL TRIAL: NCT03501043
Title: Video and Temporal Spatial Parameters Assessment of Gait After Dysport Treatment. A Pilot Study
Brief Title: Assessment of Gait After Dysport Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Alberto Esquenazi, Chairman of Physical Medicine and Rehabilitation, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5075
Record Dates: First submitted 2018-04-04; First posted 2018-04-18 (Actual); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Equinovarus; Acquired
MeSH Terms: conditions — Clubfoot | interventions — abobotulinumtoxinA

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dysport (Experimental): Subjects will receive 1000 to 1500 units of Dysport to be distributed on the basis of clinical indication to ankle plantar flexors (gastrocnemius and soleus), knee extensors and flexors, tibialis posterior and long toe flexors for one injection.
  Interventions: Drug: Dysport

INTERVENTIONS:
Drug: Dysport — Dysport 1000 to 1500 units to be distributed on the basis of clinical indication to ankle plantar flexors (gastrocnemius and soleus), knee extensors and flexors, tibialis posterior and long toe flexors.
  Other Names: abobotulinumtoxinA

SUMMARY:
This pilot study will aim to understand the potential benefit of the assessment of walking using video slow motion for muscle selection and the development of an image catalogue guide of the potential results of injection of abobotulinumtoxinA by comparing foot postures before and after injection. The objective is to evaluate the use of video assessment to improve muscle selection for the injection of botulinum toxin A to improve walking outcomes. Primary outcomes include: self-selected velocity (SSV), maximal velocity (MV) and symmetry of walking. Secondary outcomes include: passive range of motion (PROM), Modified Ashworth Scale (MAS) and the Tardieu Scale (TS). Fifteen persons post stroke or TBI over age 18 with equinovarus foot deformity who are able to ambulate will be included in the study. Dysport 1000 to 1500 units will be used to be distributed on the basis of clinical indication to ankle plantar flexors (gastrocnemius and soleus), tibialis posterior and long toe flexors. The duration of subjects' participation is 4-6 weeks.

DETAILED DESCRIPTION:
This is a prospective, single arm, non-randomized clinical study with pre-post assessment to include post-stroke and Traumatic Brain Injury (TBI) outpatients with spastic ankle / foot muscles amenable to botulinum toxin injection. Subjects must be able to walk without braces.

AbobotulinumtoxinA injection in a dose range of 500 to 1500 units one time to be distributed on the basis of clinical indication to ankle plantar flexors (gastrocnemius and soleus), knee extensors, knee flexors, tibialis posterior and long toe flexors.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged ≥ 18
* Equinovarus foot deformity appropriate for botulinum toxin treatment (naïve or non-naïve)
* Modified Ashworth Scale between 1 to 3
* Women of reproductive potential must use effective contraception for the duration of the study

Exclusion Criteria:

* Inability to walk without leg brace
* Previous surgical intervention to affected/ankle/foot
* Uncontrolled seizures
* Pregnancy or lactation
* Known allergic reactions to Dysport
* Treatment with another investigational drug or other intervention in the past 4 months
* Modified Ashworth Scale 4
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study
* Lower motor neuron disorder
* < Four months post botulinum toxin or serial casting

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Esquenazi, MD, Principal Investigator — MossRehab
Locations (1):
- MossRehab, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dysport: All Participants
Period: Overall Study
Arm/Group | Dysport
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Post-stroke and TBI outpatients with spastic ankle / foot muscles amenable to botulinum toxin injection.
Arm/Group | Dysport
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Diagnosis [Count of Participants; unit: Participants]
  TBI | 2
  Stroke | 8
Paretic Side [Count of Participants; unit: Participants]
  Left | 5
  Right | 5

OUTCOME MEASURES:

1. Primary Outcome: Self-Selected Velocity (SSV)
Description: Baseline and follow-up SSV with and without shoes. Distance covers over time at self selected pace. Larger value is better.
Time Frame: Baseline, Follow-up (4-6 weeks)
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Barefoot SSV: SSV reported in participants walking barefoot.
- Shoes SSV: SSV reported in participants walking in shoes.
Arm/Group | Barefoot SSV | Shoes SSV
Number analyzed (Participants) | 10 | 10
m/s
  Baseline | 0.41 (.31) | .48 (.27)
  Follow-up | 0.48 (.29) | 0.52 (.29)

2. Primary Outcome: Maximal Velocity
Description: Baseline and follow-up MV with and without shoes. Distance covers over time when walking as fast as possible. Larger value is better.
Time Frame: Baseline, Follow-up (4-6 weeks)
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Barefoot MV: MV reported in participants walking barefoot.
- Shoes MV: MV reported in participants walking in shoes.
Arm/Group | Barefoot MV | Shoes MV
Number analyzed (Participants) | 10 | 10
m/s
  Baseline | .59 (.48) | .71 (.41)
  Follow-up | .64 (.47) | .78 (.44)

3. Primary Outcome: Step-length at Baseline and at Follow-up (Temporal-spatial Data)
Description: Step length measured as the distance between the heel contact point of one foot and that of the other foot.
  Values are reported on the involved side. Larger values represent better outcome.
Time Frame: Baseline, Follow-up (4-6 weeks)
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Barefoot Step-Length: Step-length reported in participants walking barefoot.
- Shoes Step-Length: Step-length reported in participants walking in shoes.
Arm/Group | Barefoot Step-Length | Shoes Step-Length
Number analyzed (Participants) | 10 | 10
meters
  Baseline | .47 (.30) | .50 (.13)
  Follow-up | .50 (.12) | .51 (.14)

4. Secondary Outcome: Modified Ashworth Scale (MAS) at Baseline and at Follow-up
Description: Passive range of ankle in 1 second with knee flexed and knee extended. Scale of 0-4 (0: no increase in muscle tone; 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+:Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement); 2: More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved; 3: Considerable increase in muscle tone passive, movement difficult; 4: Affected part(s) rigid in flexion or extension.
  0-4 (Min-Max) Higher scores represents increase abnormal tone.
Time Frame: Baseline, Follow-up (4-6 weeks)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- MAS Ankle Knee Flexed: Change in ankle knee flexion MAS score
- MAS Ankle Knee Extended: Change in ankle knee extension MAS score
Arm/Group | MAS Ankle Knee Flexed | MAS Ankle Knee Extended
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 2 [1.63 to 2] | 3 [2 to 3]
  Follow-up | 1 [0.25 to 1.5] | 1 [1 to 1]

5. Secondary Outcome: Tardieu Scale (TS) at Baseline and at Follow-up
Description: Measurement of spastic response when passively ranging the ankle joint at very slow and very fast velocities with knee flexed and knee extended.
  Quality of muscle reaction (scored 0-4). 0 is no resistance to passive ROM to 4 indicating joint is immobile.
Time Frame: Baseline, Follow-up (4-6 weeks)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- TS Ankle Knee Flexed Spasticity Grade; TS Ankle Knee Extended Spasticity Grade: Participants were measured by the muscles' responses to stretch at given velocities.
Arm/Group | TS Ankle Knee Flexed Spasticity Grade | TS Ankle Knee Extended Spasticity Grade
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 3 [2 to 3] | 3 [3 to 3]
  Follow-up | 1 [1 to 1] | 1 [1 to 1]

6. Secondary Outcome: Passive Range of Motion (PROM) at Baseline and at Follow-up
Description: Normal ranges of ankle dorsiflexion 0 to 30 degrees with knee flexed. Normal ranges of dorsiflexion 0 to 15 degrees with knee extended. Higher values in dorsiflexion range represent a better outcome.
Time Frame: Baseline, Follow-up (4-6 weeks)
Population: Clinician moved the ankle at flexion or extension with no effort from the participant.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- PROM Ankle Knee Flexed: PROM measured at ankle knee flexed.
- PROM Ankle Knee Extended: PROM measured at ankle knee extended.
Arm/Group | PROM Ankle Knee Flexed | PROM Ankle Knee Extended
Number analyzed (Participants) | 10 | 10
degrees
  Baseline | 44 (13.3) | 34 (13.1)
  Follow-up | 50 (7.8) | 45.7 (9.6)

ADVERSE EVENTS:
Time Frame: Adverse event was collected at follow-up (4-6 weeks) after the baseline visit.
Groups:
- Dysport: Participants that received Dysport.
Arm/Group | Dysport
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport (N=11)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT03501043/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT03501043/Prot_SAP_001.pdf